CLINICAL TRIAL: NCT03908138
Title: RDD Versus VDD in Newly Diagnosed Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Hematology, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongPH03
Record Dates: First submitted 2019-03-28; First posted 2019-04-09 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-04

CONDITIONS: Hematologic Neoplasms; Multiple Myeloma; Efficacy; Safety
Keywords: multiple myeloma; lenalidomide
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: The patients will be randomized either receiving RDD or receiving VDD therapy.
Masking Description: no mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDD group (Active Comparator): Lenalidomide: 25mg, po, d1-21， Pegylated Liposomal Doxorubicin: 30-40mg/m2，ivgtt, d1 Dexamethasone: 20-40mg, po, d1，d8，d15，d22
  Interventions: Drug: RDD
- VDD group (Active Comparator): Bortezomib:1.3mg/m2，ih，d1，d4，d8，d11 Pegylated Liposomal Doxorubicin: 30-40mg/m2，ivgtt, d1 Dexamethasone: 20 mg, ivgtt, d1, 2, 4, 5, 8, 9, 11,12
  Interventions: Drug: VDD

INTERVENTIONS:
Drug: RDD — Lenalidomide: 25mg, po, d1-21， Pegylated Liposomal Doxorubicin: 30-40mg/m2，ivgtt, d1 Dexamethasone: 20-40mg, po, d1，d8，d15，d22
  Other Names: RDD group
  Arms: RDD group
Drug: VDD — Bortezomib:1.3mg/m2，ih，d1，d4，d8，d11 Pegylated Liposomal Doxorubicin: 30-40mg/m2，ivgtt, d1 Dexamethasone: 20 mg, ivgtt, d1, 2, 4, 5, 8, 9, 11,12
  Other Names: VDD group
  Arms: VDD group

SUMMARY:
Multiple myeloma (MM) is a common malignant hematology disease. The development of proteasome inhibitors (PIs) and immunomodulatory drugs (IMiDs) significantly improved the survival of MM patients. IMiDs have multiple effects in MM therapy. Except for direct cytotoxicity, IMiDs also play a variety of immune regulatory roles. Lenalidomide, a kind of IMiDs, was usually used in the therapy of relapsed/refractory MM. The efficacy and safety of RDD (lenalidomide, pegylated liposomal doxorubicin, dexamethasone) in newly diagnosed patients with MM still needs to be further validated.

DETAILED DESCRIPTION:
The therapy regimens of MM were very limited before 2000, mainly including VAD (vincristine, doxorubicin, dexamethasone), methylpheniram, corticosteroids and autologous stem cell transplantation (ASCT). The development of proteasome inhibitors (PIs) and immunomodulatory drugs (IMiDs) in the 2000's significantly improved the survival of MM patients. Combined chemotherapy containing new drugs has become the first-line therapy for the treatment of newly diagnosed MM patients.

In addition to direct cytotoxicity, IMiDs also play a variety of immune regulatory roles. The effects on immune system include reducing TNF-α, IL-1β, IL-6 and IL-12, increasing production of IL-2 and IFN-γ, increasing T cell initiation, enhancing the absorption of tumor antigen by dendritic cells (DCs), enhancing the efficiency of antigen presentation, inhibiting regulatory T cells (Treg), and enhancing the activity of natural killer cells (NK) and NKT cells. Lenalidomide, a kind of IMiDs, also have the effects on osteoclasts, which are important in bone disease in MM patients.

In 2006, the combination of lenalidomide and dexamethasone (RD) was approved in the United States for the treatment of relapsed/refractory MM. The RD regimen was approved for the treatment of newly diagnosed MM patients in 2015. Four lenalidomide-containing triple drug regimens were approved for the treatment of relapsed/refractory MM from 2015 to 2016. However, the application of lenalidomide-containing triple drug regimens in newly diagnosed patients with multiple myeloma needs to be further validated. Therefore, we designed the randomized controlled clinical study and aimed to compare the efficacy and safety between RDD (lenalidomide, pegylated liposomal doxorubicin, dexamethasone) and VDD (bortezomib, pegylated liposomal doxorubicin, dexamethasone) in newly diagnosed patients with MM.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of symptomatic (active) MM;
* Ages ≥18 years old, ≤65 years old;
* ECOG score: 0-2;
* Liver function: transaminase≤2.5×upper limit of normal value，bilirubin≤1.5×upper limit of normal value;
* Renal function: serum creatinine is 44-176 mmol/L;
* LVEF≥50%;
* New York Heart Association (NYHA) heart function classification is I-II grade;
* Signed informed consent.

Exclusion Criteria:

* Severe complications or severe infection;
* Severe heart disease history, including ventricular tachycardia (VT), atrial fibrillation (AF), heart block, myocardial infarction (MI), congestive heart failure (CHF), coronary heart disease patients needed therapy;
* Severe allergic constitution, or those who are allergic to or intolerant of drug composition in chemotherapy regimens; with other malignant tumors in the past 5 years;
* Patients participate in other clinical studies;
* Patients are not suitable for the study;
* Other contraindications for ASCT therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-03-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) | At 8 months
  meeting the standard IMWG response criteria (CR and VGCR) of NCCN guidelines (Version2. 2019)
partial remission (PR) | At 8 months
  meeting the standard IMWG response criteria (PR) of NCCN guidelines (Version2. 2019)

SECONDARY OUTCOMES:
Progressive free survival | At 3 months, 5 months, 8 months, 12 months, 18 months, 24 months and 36 months
  the length of time during and after the treatment of MM that a patient lives with the disease but it does not get worse
overall survival (OS) | At 3 months, 5 months, 8 months, 12 months, 18 months, 24 months and 36 months
  the percentage of MM patient who are alive after 3 years.

OTHER OUTCOMES:
Side effects | At 3 months, 5 months and 8 months
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, PhD, MD, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Department of Hematology, Provincial Hospital Affiliated to Shandong University, Jin'an, Shandong, China

IPD SHARING:
Plan to Share IPD: No